CLINICAL TRIAL: NCT01075373
Title: A Neurobiological Study on Heterogeneity of Schizophrenia: Genetic Variations and Neurobiological Differentiations
Acronym: SONPOS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Hai-Gwo Hwu, National Taiwan University Hospital
Other Study IDs: 200807021R; NSC 97-2321-B-002-041- (Other Grant/Funding Number: National Science Concil); NSC 98-2321-B-002-008- (Other Grant/Funding Number: National Science Concil)
Record Dates: First submitted 2010-02-23; First posted 2010-02-25 (Estimated); Last update posted 2010-03-08 (Estimated); Status verified 2010-02

CONDITIONS: Schizophrenia
Keywords: early stage schizophrenia; drug naïve schizophrenia; treatment response; Aripiprazole; pharmacogenetics; Disrupted-in-Schizophrenia 1 gene (DISC1); Neuregulin 1 gene (NRG1); Dopamine receptor type 2 gene (DRD2); Catechol-O-Methyltransferase gene (COMT); neurocognitive function; event-related evoked potential (ERP); Niacin skin test; plasma neurotransmitter level; plasma cytokine level; plasma signaling protein level; AKT1 protein level in the peripheral lymphocytes; 16-45 y/o; without mental retardation or epilepsy
MeSH Terms: conditions — Schizophrenia; Fibromatosis, Gingival, 2; Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Schizophrenia (SCH) is a devastating brain disorder with grave personal, family and social cost. SCH is a complex and heterogeneous (both genetic and clinical) disorder with oligogenetic endowed vulnerability risk of disease, which manifested as a clinical syndrome comprised of positive, negative and cognitive symptoms in late adolescent or young adulthood under the interaction with environmental stress. The fact that most positive psychotic symptoms can be well controlled by dopamine-blocking antipsychotics substantiates that dopamine hyperactivity is the pathophysiological model of SCH positive symptoms. This is the dopamine model of SCH.

The presence of negative and cognitive symptoms has not being fully explained by the dopamine model. The hypo-glutaminergic function was hypothesized to replace or to supplement the dopamine pathological model. The hypo-glutaminergic state was due to a neurodevelopmental disturbance in early-stage of life, and was coined as a pathophysiological mechanism of SCH.

The neurodevelopmental disturbance supports the hypo-glutamine model based on the cytoarchitecture abnormality in glutamate-pyramidal cells and reduced gray matter volume. We have found potential vulnerability genes of DISC1 and NRG1 in our Taiwanese SCH family samples. These two genes have functions on neurodevelopmental process. Besides, we, the investigators, also found two vulnerability genes of DRD2 receptor gene and COMT genes in our Taiwanese SCH families. The dopamine neurotransmission disturbance could be another pathophysiological mechanism of SCH.

With the awareness of confounding variables of antipsychotic treatment response revealed in pharmacogenetic studies, such as drug metabolism related genes and plasma HVA level, we intend to test the etiological genetic hypotheses in antipsychotic treatment response: (1) The group of neurodevelopmental etiology with risk variations in DISC1 and NRG1 genes is of poor treatment response group; (2) The group of pure hyperdopamine etiology with risk variation in DRD2 receptor and COMT genes is of good treatment group.

The potential treatment response related biomarkers, which are directly or indirectly induced by the etiological risk genetic variations, will be examined. These potential biomarkers include homovanillic acid (HVA), glutamate, serotonin, cytokines, and signaling proteins, the neurocognitive function, event-related evoked potential, Niacin skin test, and the AKT1 level in the peripheral lymphocytes.

After obtained the informed consult, we'll recruit 30 drug-naïve early schizophrenia (first episode or prodromal stage) patients for pre-treatment and post-treatment assessment on treatment response using positive and negative syndrome scale (PANSS), changes in biomarkers (including biochemical, electro-physiological and neuro-cognitive variables), and brain imaging (studies of component Project No.2 of this Integrated Program) of PET, fMRI, MRI, DSI and MRS (please refer to Project No.2) in addition to genotyping on DISC1, NRG1, DRD2 and COMT genes. The treatment agent is the dopamine stabilizing agent (aripiprazole, 15mg/day for 4 weeks) taking the advantage of dopamine activity balancing effect. Besides, we'll recruit 30 normal controls matched with age, gender, and education, who will receive genotyping and evaluations in all biomarker variables, and brain imaging studies.

In order to have adequate statistical power in the genetic analysis of 17 SNP variations in 4 vulnerability genes of DISC1, NRG1, DRD2, COMT, we'll recruit 200 more cases of schizophrenia with duration of illness less than 5 years, who have received regular clinical follow up and had good compliance on medication. The treatment response will be evaluated using PANSS. These cases will also receive all biomarker examinations and genotyping studies. For comparison, we'll also recruit 100 normal controls for study.

We'll delineate the heterogeneity issue of schizophrenia using genetic variation, neurobiological biomarkers. This study result will be beneficial for understanding pathogenesis of SCH, and for developing better treatment and prevention methods.

DETAILED DESCRIPTION:
The project will use the early stage and drug naïve schizophrenic patients as the study subjects. The specific aims are:

1. To test the hypothesis that the patient group with good antipsychotic treatment response mainly carries the risk polymorphism of DRD2 and COMT genes (the dopamine transmission genes) while the group with poor antipsychotic treatment response mainly carries the risk polymorphism of DISC1 and NRG1 genes (the neurodevelopmental genes). This association is controlled by the polymorphism of genes of drug metabolizing enzymes.
2. The good vs. poor treatment response group will have different manifestation patterns in biomarkers directly or indirectly related to neurodevelopmental or dopamine neurotransmission genes. These potential biomarkers included biochemical parameters, electrophysiological and neurocognitive indicators.
3. The good vs. poor responder group has differential changes of the response-related biomarkers comparing pre-treatment and post-treatment status in special sub-sample of the drug-naïve early schizophrenia patients.

ELIGIBILITY:
Inclusion Criteria:

* early stage schizophrenia
* drug naïve schizophrenia
* no

Exclusion Criteria:

* with mental retardation
* with epilepsy
* with alcohol or substance abuse
* with panic or depressive disorder
* not pregnant

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 16-45 y/o early stage schizophrenia
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-11 (Estimated); Study Completion 2010-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Gwo Hwu, Professor, Principal Investigator — National Taiwan University Hopsital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan